CLINICAL TRIAL: NCT00211146
Title: An Open-Label, Randomized, Parallel-Group Study to Confirm the Safety and Efficacy of Epoetin Alfa (PROCRIT) Administered Perioperatively vs. the Standard of Care in Blood Conservation in Subjects Undergoing Major Elective Spinal Surgery
Brief Title: A Study to Confirm the Safety and Efficacy of Epoetin Alfa (PROCRIT) Administered Perioperatively vs. the Standard of Care in Blood Conservation in Patients Undergoing Major Elective Spinal Surgery (SPINE Study)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: Ortho Biotech, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR004621
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2011-06-10 (Estimated); Status verified 2010-04

CONDITIONS: Anemia; Venous Thrombosis
Keywords: Anemia, erythropoetin, PROCRIT, deep vein thrombosis, thrombovascular event
MeSH Terms: conditions — Anemia; Venous Thrombosis | interventions — Epoetin Alfa

INTERVENTIONS:
Drug: epoetin alfa

SUMMARY:
This study is designed to investigate the incidence of deep vein thrombosis in patients receiving a perisurgical regimen of epoetin alfa (PROCRITÂ®) as compared to patients receiving standard of care blood conservation management.

DETAILED DESCRIPTION:
The objective of the study is to demonstrate that there is no clinically important additional risk for deep vein thrombosis (DVT) in adult spine surgery using a perisurgical regimen of epoetin alfa (PROCRIT®) versus the standard of care for blood conservation. Spine surgery was selected as the population to study because anti-coagulant therapy is not always administered in association with this surgery type. In addition, the efficacy of epoetin alfa (PROCRIT®) in protecting patients from receiving allogeneic red cell transfusion across adult spinal procedures will be studied. Patients scheduled for elective spinal surgery, who agree to participate in the study, and meet eligibility criteria will be randomly assigned to epoetin alfa (PROCRIT®) or standard of care. No perioperative anti-coagulation therapy is to be administered during the study. The study hypothesis is that there is no increased risk of DVT in patients receiving perisurgical epoetin alfa (PROCRIT®) treatment. Epoetin alfa (PROCRIT®) 600U/kg administered once per week for 3 weeks prior to surgery and on the day of surgery.

ELIGIBILITY:
Inclusion Criteria:

* Subjects scheduled for elective spinal surgery (with a minimum of 3-weeks lead time) with significant anticipated perioperative blood loss (2-4 units of blood)
* Hemoglobin >10 and < 13 g/dL at screening
* Female subjects must be post menopausal for at least one year, surgically incapable of childbearing (hysterectomy or tubal ligation), or practicing an acceptable method of birth control (e.g., hormonal contraceptives, intrauterine devices, or barrier and spermicide). The subject should continue with the same method for the duration of the study. If a female subject is practicing an acceptable method of birth control, she must have maintained her normal menstrual pattern within the three months prior to study entry
* No clinically significant abnormal hematologic or serum chemistry values. Negative serum pregnancy test for female subjects not post menopausal for at least one year or surgically incapable of childbearing (hysterectomy or tubal ligation)

Exclusion Criteria:

* No primary hematologic disease
* No clinically significant disease/dysfunction of the cardiovascular (NYHA Classification Class II-IV), neurologic (cerebral), pulmonary, endocrine, gastrointestinal, or genitourinary systems, which in the opinion of the investigator would put the subject at increased risk for a thrombovascular event, compromise the subject's ability to respond to r-HuEPO therapy, or otherwise impair their ability to participate in this study
* No history of deep vein thrombosis (DVT) or pulmonary embolism (PE)
* No subjects who are to receive perioperative pharmacologic anticoagulation (e.g., coumadin, heparin, lovenox, aspirin/ASA)
* No subjects prohibited from receiving blood transfusions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 680 (Actual)
Dates: Start 1998-04; Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
The incidence of DVT as determined by color flow duplex imaging

SECONDARY OUTCOMES:
Incidence of TVEs; Proportion of completed subjects receiving allogeneic red cell transfusions; Change in hemoglobin and hematocrit from baseline to end of study

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Derived] Stowell CP, Jones SC, Enny C, Langholff W, Leitz G. An open-label, randomized, parallel-group study of perioperative epoetin alfa versus standard of care for blood conservation in major elective spinal surgery: safety analysis. Spine (Phila Pa 1976). 2009 Nov 1;34(23):2479-85. doi: 10.1097/BRS.0b013e3181bd163f. PMID 19927096
- See also: An Open-Label, Randomized, Parallel Group Study to Confirm the Safety and Efficacy of PROCRIT (Epoetin alfa) Administered Perioperatively Versus the Standard of Care in Blood Conservation in Subjects Undergoing Major Elective Spinal Surgery — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=608&filename=CR004621_CSR.pdf